CLINICAL TRIAL: NCT05181670
Title: The Canadian Respiratory Research Network Long COVID-19 Study
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Andrea Gershon, Scientist and Respirologist, Sunnybrook Health Sciences Centre
Other Study IDs: 177755
Record Dates: First submitted 2022-01-04; First posted 2022-01-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV-2 Infection; Post-acute Sequelae of SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preliminary studies suggest that COVID-19 causes long-term lung damage, even in young, otherwise healthy people who did not need to go to hospital or the ICU.

We seek to know how common long-term lung damage after COVID-19 is, who is most affected by it and what the effects of this damage are on other important aspects of people's lives. We plan to study a large sample of people with a history of COVID-19 infection from across Canada-some who needed hospitalization but most who did not. Through online questionnaires, we will determine their respiratory symptoms, quality of life and medical history. Then we will invite them to one of our thirteen Canadian testing centres to have special, thorough breathing tests.

We hypothesize that COVID-19 leaves a significant proportion of people with measurable respiratory impairment.

The information we learn about the effect of COVID-19 on the lungs will help patients and health care providers manage it better. It will also reveal how different COVID-19 variants affect the lungs. We will use this new knowledge to write a formal guide on what respiratory monitoring and testing should be done after COVID-19 infection. This will ensure that people affected by COVID-19 get the care they need to maintain their lung health.

DETAILED DESCRIPTION:
We will prospectively recruit a representative, random sample of adult (age ≥ 18), community-dwelling patients, who have had a positive PCR test for COVID-19 infection and symptomatic infection five to 12 months previously.

This cross-sectional, observational study will have two phases:

1. Screening:

   Screening for eligibility
2. Observation Period:

   1. Online / telephone visit: All participants will complete a series of questionnaires (either online or by phone with the assistance of research personnel). In the questionnaires they will be asked about respiratory symptoms (the primary outcome), baseline participant data, burden of respiratory symptoms, overall quality of life, mental health issues as well as physical and psychological trauma from COVID-19.
   2. In-person visit: All participants will complete pulmonary function testing including oscillometry.

The study of COVID-19 infection and its long-term effects is constantly evolving. Over the course of this research study, new knowledge may become available that may lead to changes in the study's outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* Community dwelling
* First occurrence of a positive diagnostic test for SARS-CoV-2 infection (i.e., PCR or rapid antigen test, including at-home rapid antigen test) and symptomatic infection 5-12 months previously
* Consent provided
* Willing and able to go to study site for pulmonary function testing including oscillometry

Exclusion Criteria:

- Not able to communicate with our research personnel (themselves or through a translator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of respiratory post-acute sequelae of SARS-CoV-2 (PASC) and PASC | At five-12 months post positive PCR test for SARS-CoV-2 infection

SECONDARY OUTCOMES:
To determine risk factors for respiratory PASC | At five-12 months post positive PCR test for SARS-CoV-2 infection
To determine the spectrum of severity of respiratory PASC | At five-12 months post positive PCR test for SARS-CoV-2 infection
To determine objective physiologic characteristics of respiratory PASC | At five-12 months post positive PCR test for SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gershon, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (8):
- Canada (8):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec